CLINICAL TRIAL: NCT02938000
Title: E-Rehabilitation: Aerobic Resistance Training for Stroke Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB # 10926
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Stroke; Hemiplegia
Keywords: aerobic training; stroke; exercise; stroke recovery
MeSH Terms: conditions — Stroke; Hemiplegia; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Theraband group (Experimental): This group will be furnished with Thera-band, and link to exercise video, with plans for regular exercise as described previously, in addition to usual post stroke care.
  Interventions: Device: Theraband with exercise video
- Usual Care Group (Placebo Comparator): This group will have usual post stroke care, and will be advised to get regular exercise.
  Interventions: Other: usual care with advice to exercise

INTERVENTIONS:
Device: Theraband with exercise video — Theraband exercise band for resistance training
  Arms: Theraband group
Other: usual care with advice to exercise — advice to exercise
  Arms: Usual Care Group

SUMMARY:
This pilot study intends to evaluate an online exercise video rehabilitation program for stroke survivors with moderate disability compared to usual care. The intervention videos combine aerobic and resistance training using a latex resistance band, Thera band® elastic band, specifically designed for rehabilitation. This study will aim to show that for patients suffering acute ischemic stroke resulting in disability, at-home physical therapy with aerobic exercise videos will improve depression level and aerobic capacity more than usual care.

DETAILED DESCRIPTION:
Seven million Americans are stroke survivors and another four million Americans are expected to have strokes by 2030.1 Nearly 800,000 strokes occur annually and of these, 25% occur after a previous stroke or transient ischemic attack (TIA).2 Put another way, stroke recurrence affects 30% of stroke survivors.3 Given the high burden of stroke among stroke survivors, preventing recurrence is a top priority for post-stroke and post-TIA management.

Stroke survivors must cope with impairments in functioning that can range from facial droops to hemiparesis and aphasia. These physical challenges mean that even four years after stroke, 71% of survivors feel they have not completely recovered from the stroke.4 The peak oxygen cost (VO2) of participating in activities of daily living such as walking is higher in stroke survivors six months after stroke than able-bodied individuals.5,6 This increased energy cost is related to decreased cardiorespiratory reserve, changes in tissue composition, and gait deviation and asymmetry.5,6 The exhaustion point for hemiparetic stroke survivors falls within the range of aerobic fitness required to perform activities of daily living (3-5 METS [Metabolic Equivalents]).6 Small increases in aerobic capacity would therefore translate into the ability to perform activities of daily living.6

The American Heart Association (AHA) and American Stroke Association issued guidelines in 2014 recommending physical activity and exercise to improve stroke survivors' functional ability, quality of life, and morbidity of stroke recurrence.3 It is the goal of this study to improve physical activity adherence in stroke survivors and thereby improve their cardiorespiratory reserve and reduce depression. Secondary variables to be examined include functional ability, balance, blood pressure, body mass index (BMI), rates of cerebrovascular and cardiovascular events, and mortality.

Exercise-based cardiac rehabilitation post-stroke or post-TIA Cardiac rehabilitation care post-discharge for stroke survivors is not established standard of practice. Several groups have been evaluating the efficacy of comprehensive cardiac rehabilitation, as provided to patients after acute MI, in post-stroke populations. This intervention has been shown to be cost effective in post-MI care, reducing healthcare cost overall (attributed to fewer re-admissions) and per quality-adjusted life year.12 Several groups have conducted small-scale trials of cardiac rehabilitation among TIA and stroke patients with promising improvements in cardiovascular fitness outcomes.13-16 Aerobic exercise for rehabilitation after stroke has been evaluated in small randomized controlled trials.6,17

One group conducted a randomized controlled trial of a comprehensive cardiac rehabilitation program in chronic stroke patients after ischemic events.14 Their intervention was twice weekly, supervised exercise on cycle ergometers (upper or lower body) to 50-60% maximal heart rate.14 At the end of the ten-week program, subjects in the intervention arm showed significant improvements in cardiovascular fitness as measured by peak oxygen consumption (VO2) and rating of perceived exertion (RPE) after three minutes of exercise.14 Self-reported depression and anxiety scores also improved in the intervention arm, though health-related quality of life did not.14 The same group is now conducting a larger clinical trial called Cardiac Rehabilitation Adapted For Transient Ischemic Attack and Stroke (CRAFTS) expanding on the results of the earlier pilot.13,14

Another group in London, Ontario conducted a feasibility study evaluating the use of comprehensive cardiac rehabilitation (CCR) in patients within 12 months of TIA or mild, non-disabling stroke.15 In this prospective cohort study, 100 patients were enrolled and 80 patients completed the CCR with group-based or home-based progressive aerobic training for six months.15 Diet counseling in individual or group-based sessions emphasized the Mediterranean diet.15 Patients were screened for depression and referred to a psychologist for anxiety, depression, and smoking cessation as needed.15 Medications were optimized to meet AHA recommendations regarding use of aspirin or anti-platelet agent, angiotensin converting enzyme inhibitor, statin, and blood pressure management with diuretic.15 The results of the feasibility study were promising with improvements in cardiopulmonary fitness, blood lipid profile, BMI, weight, waist circumference, smoking status, and Duke Treadmill Score.15 Although the study was not powered to evaluate morbidity of stroke/TIA and mortality, the recurrence of stroke was 0% among patients who completed intake/outtake and 4.6% including patients who left CCR.15

A third study, PREVENT, is a randomized controlled trial out of Nova Scotia, Canada currently enrolling patients post-TIA or non-disabling stroke to evaluate a program of rehabilitative exercise and education in improving risk factors.16 The trial aims to randomize 250 patients to control (usual care) or to a 12-week comprehensive rehabilitation program comprising group- and home-based exercise with aerobic and resistance training and weekly education classes.16 Primary outcomes to be measured include lipid profile, blood pressure, waist circumference, fasting glucose, and hemoglobin A1c; secondary outcomes to be assessed are exercise capacity, walking endurance, cognitive function, depression, health-related quality of life, and physical activity.16 The trial was not powered to evaluate the effectiveness of the intervention in preventing morbidity of stroke/TIA/cardiac events.16

AHA Recommendation In 2014, American Heart Association (AHA)/American Stroke Association released recommendations regarding physical activity in stroke survivors.3 Prior to starting, a pre-exercise physical evaluation including electrocardiogram (ECG), heart rate monitoring, and graded exercise testing. Recommended exercise is aerobic cardiovascular exercise 3-5 times weekly for 20-60 minutes; aerobic activity should achieve 40-70% peak O2 or heart rate maximum.3 Additional exercise in resistance training two to three days weekly is also recommended.

The proposed intervention differs from these studies in that it involves a one-way communication via streaming video in addition to case management follow-up phone calls. To our knowledge, the efficacy of this tele-intervention has not been reported previously.

Thera-band® elastic bands Thera band® elastic bands (The Hygienic Corporation, Akron, Ohio) are versatile exercise training tools used primarily to provide graded resistance during strength training.22 They have been used in home-based resistance training for stroke rehabilitation with improvement in strength, gait speed, and functional ability.22 Combined with aerobic activity, strength training of hip flexors, extensors, and abductors improved gait speeds between 3.6-12.6 meters/minute in ambulatory stroke survivors after ten weeks of intervention.22-24 A small study (sponsored by the manufacturer of Thera band®) found using Thera band® elastic band is comparable to using resistance-training machines in activating exercised muscles, as demonstrated by electromyography (EMG).25 Community-based training with physiotherapists guiding stroke survivors in the use of Thera band® elastic bands for resistance training over 16 weeks improves balance and strength.26

In addition to providing resistance, Thera band® can be used to assist stroke survivors in dorsiflexion during gait training. Patients who received gait training using Thera band® showed faster improvement in mobility than usual care.27

A guided, community-based model is the most representative of e-rehabilitation. Strength and gait improvements are comparable in supervised and unsupervised resistance training in stroke survivors.23 This study's recorded exercise videos are intended to visually demonstrate aerobic resistance training to community-dwelling patients. Although the patients will remain unsupervised, exercise sessions will be entirely guided by a trained exercise physiologist.

This pilot, randomized, controlled, double-blinded study will compare a comprehensive lifestyle and exercise rehabilitation intervention to usual care in patients after acute stroke. The investigators of this study intend to evaluate an online exercise video rehabilitation program for stroke survivors with moderate disability compared to usual care. The intervention videos combine aerobic and resistance training using a latex resistance band, Thera band® elastic band, specifically designed for rehabilitation.

The proposed study will be performed at the Kaiser Permanente (KP) San Diego Medical Center. Kaiser Permanente patients that are admitted with acute ischemic stroke, resulting in moderate disability, in the prior two weeks to enrollment range will be recruited in the medical center. Patients will be directly offered participation in the study by the principal investigator, at the time of hospital admission to the KP San Diego Medical Center with ischemic stroke. For patients interested in participating in the trial, screening based on written inclusion and exclusion criteria will be done by reviewing patient information in the electronic medical record system. If patient meets initial eligibility criteria, they will be notified by telephone.

As part of usual care, all enrolled patients will have an initial study visit included within their post-hospital discharge follow-up visit. Informed consent will be obtained at this time, as well as subsequent collection of baseline data, including vital signs, social and medical history, demographic variables, and questionnaire response items.

All patients will have an appointment at Positive Choice within two weeks of the initial visit for education training, further testing (aerobic capacity measures), and distribution of Thera bands to the intervention group. Within the subsequent week patients and family in the intervention arm will receive an educational outreach call which will include medication reconciliation and adherence, dietary adjustments, smoking cessation, physical activity, depression education, as well as how to access the physical therapy videos online. Videos are 20-30 minutes with combination of aerobic and resistance training to be done in seated positions.

Study staff will call patients 1 week after the aforementioned educational phone call to offer encouragement, ask about progress, and answer any questions the patient may have regarding the videos. To control patients, the call will be a brief reminder to continue to adhere to medical therapy. Study staff will also call all enrolled patients to screen for depression at 4-week intervals, and to ensure coordination for depression treatment with primary care physician. Investigator will perform physical exam including NIH stroke scale at the completion of prescribed therapy. At this time, patient will be advised to continue physical activity with videos as part of AHA recommendation.

The outcome status (in terms of toxicity, response, reason off study, progression, and survival) of all eligible patients will be reported. All eligible patients who begin treatment will be included in the analysis of survival and time-to-failure. The primary outcomes of this study are the impact on the depression scores and cardiorespiratory reserve change of stroke survivors as a result of the intervention videos combined with aerobic and resistance training using a latex resistance bands. Additional outcomes of this study are measurement of potential changes in body mass index (BMI), blood pressure (BP), hemoglobin A1c (HbA1c), functional status, balance, incidence of cardiovascular and cerebrovascular events, as well as adherence to exercise program.

ELIGIBILITY:
Inclusion Criteria:

* acute ischemic stroke within 2 weeks of enrollment

Exclusion Criteria:

* unstable coronary artery disease, oxygen dependent, with oxygen saturation less than 92% on room air, unable to perform peak oxygen consumption testing, musculoskeletal disease limiting exercise performance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-08; Primary Completion 2017-03 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
VO2: aerobic capacity measurement with peak VO2 using 6 minute walk test | 12 weeks

SECONDARY OUTCOMES:
Berg Balance Score | 12 weeks
  standardized questionnaire to assess balance difficulty following stroke.
adherence to exercise program, interventional group only | 12 weeks
  participants will be asked how many exercise sessions they have completed in the time frame.
Patient Health Questionnaire - 9 (PHQ 9) | 12 weeks
  standardized assessment for depression following stroke

CONTACTS AND LOCATIONS:
Overall Officials: William P Neil, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Soliman EZ, Sorlie PD, Sotoodehnia N, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2012 update: a report from the American Heart Association. Circulation. 2012 Jan 3;125(1):e2-e220. doi: 10.1161/CIR.0b013e31823ac046. Epub 2011 Dec 15. No abstract available. PMID 22179539
- [Background] Furie KL, Kasner SE, Adams RJ, Albers GW, Bush RL, Fagan SC, Halperin JL, Johnston SC, Katzan I, Kernan WN, Mitchell PH, Ovbiagele B, Palesch YY, Sacco RL, Schwamm LH, Wassertheil-Smoller S, Turan TN, Wentworth D; American Heart Association Stroke Council, Council on Cardiovascular Nursing, Council on Clinical Cardiology, and Interdisciplinary Council on Quality of Care and Outcomes Research. Guidelines for the prevention of stroke in patients with stroke or transient ischemic attack: a guideline for healthcare professionals from the american heart association/american stroke association. Stroke. 2011 Jan;42(1):227-76. doi: 10.1161/STR.0b013e3181f7d043. Epub 2010 Oct 21. PMID 20966421
- [Background] Billinger SA, Arena R, Bernhardt J, Eng JJ, Franklin BA, Johnson CM, MacKay-Lyons M, Macko RF, Mead GE, Roth EJ, Shaughnessy M, Tang A; American Heart Association Stroke Council; Council on Cardiovascular and Stroke Nursing; Council on Lifestyle and Cardiometabolic Health; Council on Epidemiology and Prevention; Council on Clinical Cardiology. Physical activity and exercise recommendations for stroke survivors: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2014 Aug;45(8):2532-53. doi: 10.1161/STR.0000000000000022. Epub 2014 May 20. PMID 24846875
- [Background] Gadidi V, Katz-Leurer M, Carmeli E, Bornstein NM. Long-term outcome poststroke: predictors of activity limitation and participation restriction. Arch Phys Med Rehabil. 2011 Nov;92(11):1802-8. doi: 10.1016/j.apmr.2011.06.014. PMID 22032214
- [Background] Danielsson A, Willen C, Sunnerhagen KS. Measurement of energy cost by the physiological cost index in walking after stroke. Arch Phys Med Rehabil. 2007 Oct;88(10):1298-303. doi: 10.1016/j.apmr.2007.06.760. PMID 17908572
- [Background] Ivey FM, Hafer-Macko CE, Macko RF. Exercise rehabilitation after stroke. NeuroRx. 2006 Oct;3(4):439-50. doi: 10.1016/j.nurx.2006.07.011. PMID 17012057
- [Background] Heran BS, Chen JM, Ebrahim S, Moxham T, Oldridge N, Rees K, Thompson DR, Taylor RS. Exercise-based cardiac rehabilitation for coronary heart disease. Cochrane Database Syst Rev. 2011 Jul 6;(7):CD001800. doi: 10.1002/14651858.CD001800.pub2. PMID 21735386
- [Background] Lawler PR, Filion KB, Eisenberg MJ. Efficacy of exercise-based cardiac rehabilitation post-myocardial infarction: a systematic review and meta-analysis of randomized controlled trials. Am Heart J. 2011 Oct;162(4):571-584.e2. doi: 10.1016/j.ahj.2011.07.017. Epub 2011 Sep 3. PMID 21982647
- [Background] Suaya JA, Shepard DS, Normand SL, Ades PA, Prottas J, Stason WB. Use of cardiac rehabilitation by Medicare beneficiaries after myocardial infarction or coronary bypass surgery. Circulation. 2007 Oct 9;116(15):1653-62. doi: 10.1161/CIRCULATIONAHA.107.701466. Epub 2007 Sep 24. PMID 17893274
- [Background] McCarthy D, Mueller K, Wrenn J. Kaiser Permanente: Bridging the Quality Divide with Integrated Practice, Group Accountability, and Health Information Technology2009.
- [Background] Sandhoff BG, Kuca S, Rasmussen J, Merenich JA. Collaborative cardiac care service: a multidisciplinary approach to caring for patients with coronary artery disease. Perm J. 2008 Summer;12(3):4-11. doi: 10.7812/TPP/08-007. PMID 21331203
- [Background] Yu CM, Lau CP, Chau J, McGhee S, Kong SL, Cheung BM, Li LS. A short course of cardiac rehabilitation program is highly cost effective in improving long-term quality of life in patients with recent myocardial infarction or percutaneous coronary intervention. Arch Phys Med Rehabil. 2004 Dec;85(12):1915-22. doi: 10.1016/j.apmr.2004.05.010. PMID 15605326
- [Background] Lennon O, Blake C. Cardiac rehabilitation adapted to transient ischaemic attack and stroke (CRAFTS): a randomised controlled trial. BMC Neurol. 2009 Feb 23;9:9. doi: 10.1186/1471-2377-9-9. PMID 19236691
- [Background] Lennon O, Carey A, Gaffney N, Stephenson J, Blake C. A pilot randomized controlled trial to evaluate the benefit of the cardiac rehabilitation paradigm for the non-acute ischaemic stroke population. Clin Rehabil. 2008 Feb;22(2):125-33. doi: 10.1177/0269215507081580. PMID 18212034
- [Background] Prior PL, Hachinski V, Unsworth K, Chan R, Mytka S, O'Callaghan C, Suskin N. Comprehensive cardiac rehabilitation for secondary prevention after transient ischemic attack or mild stroke: I: feasibility and risk factors. Stroke. 2011 Nov;42(11):3207-13. doi: 10.1161/STROKEAHA.111.620187. Epub 2011 Sep 22. PMID 21940961
- [Background] MacKay-Lyons M, Gubitz G, Giacomantonio N, Wightman H, Marsters D, Thompson K, Blanchard C, Eskes G, Thornton M. Program of rehabilitative exercise and education to avert vascular events after non-disabling stroke or transient ischemic attack (PREVENT Trial): a multi-centred, randomised controlled trial. BMC Neurol. 2010 Dec 8;10:122. doi: 10.1186/1471-2377-10-122. PMID 21143864
- [Background] Pang MY, Eng JJ, Dawson AS, Gylfadottir S. The use of aerobic exercise training in improving aerobic capacity in individuals with stroke: a meta-analysis. Clin Rehabil. 2006 Feb;20(2):97-111. doi: 10.1191/0269215506cr926oa. PMID 16541930
- [Background] Williams LS, Kroenke K, Bakas T, Plue LD, Brizendine E, Tu W, Hendrie H. Care management of poststroke depression: a randomized, controlled trial. Stroke. 2007 Mar;38(3):998-1003. doi: 10.1161/01.STR.0000257319.14023.61. Epub 2007 Feb 15. PMID 17303771
- [Background] Chollet F, Tardy J, Albucher JF, Thalamas C, Berard E, Lamy C, Bejot Y, Deltour S, Jaillard A, Niclot P, Guillon B, Moulin T, Marque P, Pariente J, Arnaud C, Loubinoux I. Fluoxetine for motor recovery after acute ischaemic stroke (FLAME): a randomised placebo-controlled trial. Lancet Neurol. 2011 Feb;10(2):123-30. doi: 10.1016/S1474-4422(10)70314-8. Epub 2011 Jan 7. PMID 21216670
- [Background] Laver KE, Schoene D, Crotty M, George S, Lannin NA, Sherrington C. Telerehabilitation services for stroke. Cochrane Database Syst Rev. 2013 Dec 16;2013(12):CD010255. doi: 10.1002/14651858.CD010255.pub2. PMID 24338496
- [Background] Lysack C, Dama M, Neufeld S, Andreassi E. A compliance and satisfaction with home exercise: a comparison of computer-assisted video instruction and routine rehabilitation practice. J Allied Health. 2005 Summer;34(2):76-82. PMID 16032913
- [Background] Duncan P, Richards L, Wallace D, Stoker-Yates J, Pohl P, Luchies C, Ogle A, Studenski S. A randomized, controlled pilot study of a home-based exercise program for individuals with mild and moderate stroke. Stroke. 1998 Oct;29(10):2055-60. doi: 10.1161/01.str.29.10.2055. PMID 9756581
- [Background] Olney SJ, Nymark J, Brouwer B, Culham E, Day A, Heard J, Henderson M, Parvataneni K. A randomized controlled trial of supervised versus unsupervised exercise programs for ambulatory stroke survivors. Stroke. 2006 Feb;37(2):476-81. doi: 10.1161/01.STR.0000199061.85897.b7. Epub 2006 Jan 12. PMID 16410482
- [Background] Teixeira-Salmela LF, Olney SJ, Nadeau S, Brouwer B. Muscle strengthening and physical conditioning to reduce impairment and disability in chronic stroke survivors. Arch Phys Med Rehabil. 1999 Oct;80(10):1211-8. doi: 10.1016/s0003-9993(99)90018-7. PMID 10527076
- [Background] Andersen LL. Muscle activity during rehab exercises with Thera-band vs machine exercise. Proceedings of the 16th TRAC meeting; 2014 August 6-8, 2014; Park City, Utah. p. 16.
- [Background] Cramp MC, Greenwood RJ, Gill M, Lehmann A, Rothwell JC, Scott OM. Effectiveness of a community-based low intensity exercise programme for ambulatory stroke survivors. Disabil Rehabil. 2010;32(3):239-47. doi: 10.3109/09638280903095916. PMID 20001830
- [Background] Patil P, Rao S. Effects of Thera-Band(R) elastic resistance-assisted gait training in stroke patients: a pilot study. Eur J Phys Rehabil Med. 2011 Sep;47(3):427-33. Epub 2011 May 10. PMID 21555984
- [Background] Drew-Nord DC, Myers J, Nord SR, Oka RK, Hong O, Froelicher ES. Accuracy of peak VO2 assessments in career firefighters. J Occup Med Toxicol. 2011 Sep 25;6(1):25. doi: 10.1186/1745-6673-6-25. PMID 21943154
- [Background] Jette M, Sidney K, Blumchen G. Metabolic equivalents (METS) in exercise testing, exercise prescription, and evaluation of functional capacity. Clin Cardiol. 1990 Aug;13(8):555-65. doi: 10.1002/clc.4960130809. PMID 2204507